CLINICAL TRIAL: NCT03201705
Title: A Novel Approach in Spinal Cord Stimulation: a Combination of Burst and Tonic Waveforms.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massimo Innamorato (Other)
Responsible Party: Sponsor-Investigator, Massimo Innamorato, Director, Ospedale Santa Maria delle Croci
Organization: Ospedale Santa Maria delle Croci (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TONIC+BURST
Record Dates: First submitted 2017-06-16; First posted 2017-06-28 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Failed Back Surgery Syndrome; Spinal Cord Stimulation; Pain Management; Implantable Neurostimulator
MeSH Terms: conditions — Failed Back Surgery Syndrome; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory neuropathic leg and low back pain (Experimental): Patients with refractory neuropathic leg and low back pain as result of FBSS will be enrolled in the study and receive electrocatheter implant. Then, they will be observed for a two-weeks trial period in which the efficacy of the stimulation and the compliance of the patient is evaluated. During this trial a Tonic wave stimulation is administered by the external generator. After the trial, the definitive generator will be implanted. Tonic stimulation will be selected as wave form for four weeks. After this period, the stimulation will be switched into the combined waveform for 30 days. At the end of the study period, the final waveform setting of the SCS will be in accord with the patient's stimulation preference.
  Interventions: Device: Burst + Tonic

INTERVENTIONS:
Device: Burst + Tonic — Patients fulfilling the inclusion criteria will be enrolled in the study and receive electrocatheter implant (Precision Spectra system, Boston Scientific). Then, they will be observed for a two-weeks trial period in which the efficacy of the stimulation and the compliance of the patient is evaluated. During this trial a Tonic wave stimulation is administered by the external generator. After the trial, the definitive generator will be implanted. Tonic stimulation will be selected as wave form for four weeks. After this period, the stimulation will be switched into the combined waveform for 30 days. At the end of the study period, the final waveform setting of the SCS will be in accord with the patient's stimulation preference.

SUMMARY:
Spinal Cord Stimulation (SCS) has been a well-established treatment for chronic neuropathic pain in Failed Back Surgery Syndrome with associated legs and/or low back pain. The waves used in Spinal Cord Stimulation are mainly Tonic or Burst. Both Tonic and Burst stimulation offer neuropathic pain suppression, with slightly superiority of the Burst wave for the FBSS. The aim of our study is to evaluate the efficacy of a new stimulation paradigm with the combination of the two wave forms.

DETAILED DESCRIPTION:
Spinal Cord Stimulation (SCS) has been a well-established treatment for chronic neuropathic pain for decades. One of the most general indication for SCS is Failed Back Surgery Syndrome with associated legs and/or low back pain.

Conventional low frequency neurostimulation is applied with a tonic wave shape (pulse width is usually 300 to 500 μsec, amplitude 2 to 5 mA, and frequency 40 to 50 Hz); this kind of stimulation produces a perceptible paraesthesias in the area of stimulation "covering" the region of pain. Further development in waves of stimulation during the recent years led to new paradigms of sub-perception stimulation like "Burst" stimulation that has characteristics of a cluster of waves with higher frequency.

The efficacy of these two wave forms has been demonstrated by different authors. Both Tonic and Burst stimulation offer neuropathic pain suppression, with slightly superiority of the Burst wave for the FBSS.

Recent advances in technology of the implantable devices for spinal cord stimulation led to the possibility to combine the two stimulation waves described allowing the design of a possible new paradigm of stimulation. The Tonic and Burst wave can be combined to stimulate the same pain area using the same configuration otherwise they can be programmed to stimulate two different pain areas with two different configurations. Both burst and tonic waveforms paradigms can be customized according to patients' need. The characteristics of this combined stimulation wave in terms of efficacy, non inferiority, energy consumption, and patient satisfaction are unknown.

The primary objective of this trial is to compare pain suppressive effect of Low Frequency "Tonic Wave" versus Low Frequency Combined "Burst and Tonic Wave" for Spinal Cord Stimulation in subjects with refractory neuropathic leg and low back pain as result of FBSS.

Patients fulfilling the inclusion criteria will be enrolled in the study and receive electrocatheter implant. Then, they will be observed for a two-weeks trial period in which the efficacy of the stimulation and the compliance of the patient is evaluated. During this trial a Tonic wave stimulation is administered by the external generator. After this trial, the definitive generator will be implanted. Two weeks of Tonic stimulation will follow the surgery to avoid any interference of the pain measurement with the surgical pain. After this two weeks period, the stimulation will be switched into the combined waveform for 15 days. At the end of the study period, the final waveform setting of the SCS will be in accord with the patient's stimulation preference.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, persistent, refractory, low back pain as a result of spinal surgery
* Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and minimally interventional pain procedures for chronic pain
* Pain radiating in the leg, following segments L4 and/or L5 and/or S1 for at least 6 months
* Minimum baseline pain intensity as assessed by VAS of ≥ 50mm on 100mm scale in the primary pain area
* Subject is able and willing to provide informed consent
* Subject is able and willing to comply with the protocol and follow-up schedule

Exclusion Criteria:

* Back pain component of more than 20% or VAS > 40mm on 100mm scale
* Bilateral limb pain
* Subjects with a previous SCS implantation
* Changes in pain medication in the 2 months preceding the trial period
* Expected inability of subjects to correctly operate the neurostimulation system
* Presence of any other clinically significant or disabling chronic pain condition (eg. hip arthrosis, rheumatoid arthritis, fibromyalgia, etc.)
* History of coagulation disorders, lupus erythematosus, diabetes mellitus
* Symptoms or proof of any malignant disease
* Current use of medicines affecting coagulation which cannot be temporarily stopped
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator
* Life expectancy of less than 1 year
* Existing or planned pregnancy in the trial period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Suppression | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Pain suppression by "Tonic" and "Burst+Tonic" waves Spinal Cord Stimulation, in relation at measure previous of implant, expressed with Numerical Rate Scale (NRS)

SECONDARY OUTCOMES:
Change in quality of Life | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Oswestry Disability Index
Change in energy use of the battery | 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Energy use index (0-10): Software calculated index indicating energy consumption of the device in relation with stimulation parameters
Change in halving the pain | 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Percentage of subjects with 50% reduction in pain
Change in use of rescue medication | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Number of times in which the patient required rescue medication in a period
Change in number of stimulation adjustments | 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Number of amplitude adjustments in stimulation period
Change in discomfort due to stimulation | 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Question: are the paresthesia in the limbs acceptable? Yes/No
Change in disability | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Oswestry Disability Index
Change in subject's satisfaction | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Oswestry Disability Index
Change in social life | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Oswestry Disability Index
Change in sleep pattern | Baseline (pre intervention), 15 days and 30 days of Tonic Stimulation, 15 days and 30 days of Combined Stimulation
  Oswestry Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Innamorato, MD, Study Director — Ospedale Santa Maria delle Croci

IPD SHARING:
Plan to Share IPD: Undecided